CLINICAL TRIAL: NCT04344444
Title: Treatment in Patients With Suspected or Confirmed COVID-19 With Early Moderate or Severe Disease: A Randomized Clinical Trial
Brief Title: Treatment in Patients With Suspected or Confirmed COVID-19 With Early Moderate or Severe Disease
Acronym: RCT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy data from other studies
Sponsor: LCMC Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID 2020-001
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (No Intervention): Supportive Care only
- Arm B (Experimental): Hydroxychloroquine 400 mg po bid on Day 1 Hydroxychloroquine 200 mg po bid Days 2 through 5
  Interventions: Drug: Hydroxychloroquine
- Arm C (Experimental): Hydroxychloroquine as in Arm B AND Azithromycin 500 mg po on Day 1 Azithromycin 250 mg po days 2 through 5
  Interventions: Drug: Hydroxychloroquine; Drug: Azithromycin

INTERVENTIONS:
Drug: Hydroxychloroquine — tablets provided as described in Arm B
  Arms: Arm B; Arm C
Drug: Azithromycin — tablets provided as described in Arm C
  Arms: Arm C

SUMMARY:
This study proposes to evaluate clinical outcomes and viral load in COVID-19 infected patients with early moderate and severe disease admitted to the hospital and randomized to one of three arms. Patients will be randomized to supportive care, OR hydroxychloroquine alone, OR hydroxychloroquine and azithromycin.

DETAILED DESCRIPTION:
This is a phase 3 study.

Primary Objective:

• To evaluate clinical outcomes in patients with suspected or confirmed COVID-19 with early moderate to severe disease in a randomized controlled trial.

Secondary Objectives:

* To evaluate quantitative viral load over time
* To evaluate length of hospital stay and days in ICU
* To evaluate toxicity of the treatment options
* To evaluate rate of readmission after hospital discharge
* To evaluate duration of clinical symptoms

Arm A:

Control Arm - Supportive Care Only

Arm B:

Hydroxychloroquine 400 mg po bid on Day 1 Hydroxychloroquine 200 mg po bid Days 2 through 5

Arm C:

Hydroxychloroquine as in Arm B AND Azithromycin 500 mg po on Day 1 Azithromycin 250 mg po days 2 through 5

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Positive SARS-CoV-2 testing or consistent clinical syndrome (based on clinical picture e.g. characteristic infiltrates on chest x-ray, laboratory findings, and with agreement by two physicians) in patients under investigation (PUIs).
* Onset of symptoms < 7 days from date of enrollment
* Oxygen saturation of >94% on room air with defined risk factors (Table 1) consistent with moderate disease OR oxygen saturation of < 94% on room air consistent with severe disease
* Ability and willingness to comply with study procedures

Exclusion Criteria:

* QTc greater than 450 milliseconds on screening EKG
* Pregnant or lactating women
* Inability to take oral pills or inability to use a feeding tube
* Inability to obtain informed consent either from the patient or from the next of kin if patient is incapacitated. For the purpose of this study obtaining a verbal consent from a family member on the phone with a witness will be considered acceptable since there is a 'no visitor' policy in force at hospitals.
* Patients requiring ICU level care
* use of azithromycin or hydroxychloroquine within 30 days prior to admission

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Most severe outcome | 5 days
  ordinal outcome of most severe a patient experienced after inpatient admission

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Clement, MD, Principal Investigator — LSUHSC/UMCNO
Locations (1):
- University Medical Center New Orleans, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT04344444/ICF_000.pdf